CLINICAL TRIAL: NCT03039283
Title: Retrospective Post-market Hearing Performance Outcome in a Cohort of CI532 Recipients
Brief Title: Retrospective CI532 Hearing Performance
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL5661
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-07

CONDITIONS: Hearing Loss
Keywords: Moderate to profound sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nucleus CI532 cochlear implant
  Interventions: Device: Nucleus CI532 cochlear implant

INTERVENTIONS:
Device: Nucleus CI532 cochlear implant — Retrospective study of the commercial CI532 cochlear implant

SUMMARY:
The aim of this retrospective study is to collect and assess hearing performance data that have been measured by five clinics in Germany as part of their clinical routine in recipients implanted with a commercial CI532.

DETAILED DESCRIPTION:
Speech understanding data in quiet and in noise and aided and unaided thresholds, medical history, anomalies in terms of electrode placement are collected through an eCRF. Recipient's device characteristics are collected through cdx files. Surgeon handling and usability of CI532 are collected through paper questionnaire.

The retrospective study is aimed at collection of data for CI532 recipients who have routine hearing measures at pre-implant and post-implant intervals in their medical records.

Patients are approached for study participation by the caring clinician on a consecutive and voluntary basis and on condition of signing the patient informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Ability to conduct adult hearing performance test material
* Good German language skills to assess clinical hearing performance
* CI532 recipients assessed via routine clinical measurements at pre implant, and post implant intervals with available data records in hospital files.
* Patients that have read, understood and signed the patient informed consent.

Exclusion Criteria:

* Recipients that have participated in the CLTD5446 study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with a commercial CI532 and for which clinical routine hearing measures data are available in their medical records.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Volckaerts, PhD, Study Director — Cochlear
Locations (5):
- Germany (5):
  - Universitätsklinik für Hals-, Nasen- und Ohrenheilkunde, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Hals-Nasen-Ohren-Klinik, Erlangen, Bavaria
  - Klinikum der J. W. Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Deutsches HörZentrum Hannover der HNO-Klinik der MHH, Hanover, Lower Saxony
  - : Klinik für Hals-, Nasen-, Ohrenheilkunde, Kopf- und Halschirurgie, Kiel, Schleswig-Holstein

REFERENCES:
- [Background] Holden LK, Finley CC, Firszt JB, Holden TA, Brenner C, Potts LG, Gotter BD, Vanderhoof SS, Mispagel K, Heydebrand G, Skinner MW. Factors affecting open-set word recognition in adults with cochlear implants. Ear Hear. 2013 May-Jun;34(3):342-60. doi: 10.1097/AUD.0b013e3182741aa7. PMID 23348845
- [Background] Dowell RC, Hollow R, Winton E. Outcomes for cochlear implant users with significant residual hearing: implications for selection criteria in children. Arch Otolaryngol Head Neck Surg. 2004 May;130(5):575-81. doi: 10.1001/archotol.130.5.575. PMID 15148179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 162 participants were recruited in five German centres from March 2017 to August 2018
Period: Overall Study
Arm/Group | Nucleus CI532 Cochlear Implant
Started | 162
Completed | 160
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: 159 participants were analyzed (two protocol deviations and one participant asked to be withdrawn retrospectively)
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 86
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 159

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-operative (Daily Listening Condition) Baseline Speech Understanding in Quiet at 6 Months Post-operative (Best Aided Conditions).
Description: Is tested using the centre's clinical routine speech tests. Participants are listening in their normal hearing configuration: often with acoustic hearing aids in both ears preoperatively, an implant in one ear and hearing aid in the opposite, or using two implants, one in each ear postoperatively. All centres used Freiburger German monosyllable lists. Recorded lists of everyday words are presented to participants at 65 dB SPL (loud conversational speech level) from loudspeakers and participants repeat back what they hear. Lists are scored as a percentage correct words, with two lists being used per condition to represent speech understanding in quiet.
Time Frame: pre-operatively and at 6 months post-operatively
Population: 49 participants with routine speech understanding data available at pre-op and 6 months were analysed.
Measure: Mean (Standard Deviation); unit: Percent correct
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 49
Percent correct | 26.1 (26.7)

2. Primary Outcome: Change From Pre-operative (Daily Listening Condition) Baseline Speech Understanding in Noise at 6 Months Post-operative (Best Aided Conditions).
Description: Is tested using the centre's clinical routine speech tests. Participants are listening in their normal hearing configuration: often with acoustic hearing aids in both ears preoperatively, an implant in one ear and hearing aid in the opposite, or using two implants, one in each ear postoperatively. Centres used different types of speech in noise testing. Lists of sentences were presented in competing background noise. An adaptive procedure is used such that after each sentence is presented the speech level is decreased if >50% of the words are correctly repeated in the sentence, or increased if otherwise. The test result is the mean signal-to-noise ratio of the last eight presentations. An average of two lists is used as the result representing the signal-to-noise ratio that gives 50% sentence understanding.
Time Frame: pre-operatively and at 6 months post-operatively
Population: 15 participants with routine speech understanding data in noise available at pre-op and at 6 months were analyzed.
Measure: Mean (Standard Deviation); unit: Speech Recognition Threshold in decibels
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 15
Speech Recognition Threshold in decibels | -5.5 (11.2)

3. Primary Outcome: Percentage of Participants Showing Post-operative Improvement in the Ipsilateral Ear in Quiet.
Description: Is tested using the centre's clinical routine speech. Participants are listening using only the ear which was treated using hearing aid preoperatively and the implant postoperatively. All centres used Freiburger German monosyllable lists. Recorded lists of everyday words are presented to participants at 65 dB SPL (loud conversational speech level) from loudspeakers and participants repeat back what they hear. Lists are scored as a percentage correct words, with two lists being used per condition to represent speech understanding in quiet.
Time Frame: pre-operatively and at 6 months post-operatively
Population: 99 of the 159 participants had pre-operative and 6-month post-operative data available in the ipsilateral condition to compare.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 99
Percentage of participants | 96 [90 to 98.9]

4. Primary Outcome: Percentage of Participants Showing Post-operative Improvement in Best Aided Condition in Quiet
Description: Is tested using the centre's clinical routine speech. Participants are listening in their normal hearing configuration: often with acoustic hearing aids in both ears preoperatively, an implant in one ear and hearing aid in the opposite, or using two implants, one in each ear postoperatively. All centres used Freiburger German monosyllable lists. Recorded lists of everyday words are presented to participants at 65 dB SPL (loud conversational speech level) from loudspeakers and participants repeat back what they hear. Lists are scored as a percentage correct words, with two lists being used per condition to represent speech understanding in quiet.
Time Frame: Pre-operatively and at 6 months post-operatively
Population: 60 of the 159 participants had pre-operative and 6-month post-operative data available in the best aided condition to compare.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 60
Percentage of participants | 73.3 [60 to 84]

5. Primary Outcome: Percentage of Participants Showing Post-operative Improvement in the Ipsilateral Ear in Noise.
Description: Is tested using the centre's clinical routine speech. Participants are listening using only the ear which was treated using hearing aid preoperatively and the implant postoperatively. Centres used different types of speech in noise testing. Lists of sentences were presented in competing background noise. In some cases the noise level was fixed at 10 dB signal-to-noise ratio, and the percentage of words correctly repeated was recorded (over two lists). Alternatively, an adaptive procedure is used such that after each sentence is presented the speech level is decreased if >50% of the words are correctly repeated in the sentence, or increased if otherwise. The test result is the mean signal-to-noise ratio of the last eight presentations. An average of two lists is used as the result representing the signal-to-noise ratio that gives 50% sentence understanding.
Time Frame: Pre-operatively and at 6 months post-operatively
Population: 36 of the 159 participants had pre-operative and 6-month post-operative data available in the ipsilateral condition to compare.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 36
Percentage of participants | 67 [49 to 81]

6. Primary Outcome: Percentage of Participants Showing Post-operative Improvement in Best Aided Condition in Noise.
Description: Is tested using the centre's clinical routine speech. Participants are listening in their normal hearing configuration: often with acoustic hearing aids in both ears preoperatively, an implant in one ear and hearing aid in the opposite, or using two implants, one in each ear postoperatively. Centres used different types of speech in noise testing. Lists of sentences were presented in competing background noise. In some cases the noise level was fixed at 10 dB signal-to-noise ratio, and the percentage of words correctly repeated was recorded (over two lists). Alternatively, an adaptive procedure is used such that after each sentence is presented the speech level is decreased if >50% of the words are correctly repeated in the sentence, or increased if otherwise. The test result is the mean signal-to-noise ratio of the last eight presentations. An average of two lists is used as the result representing the signal-to-noise ratio that gives 50% sentence understanding.
Time Frame: Pre-operatively and at 6 months post-operatively
Population: 4 of the 159 participants had pre-operative and 6-month post-operative data available in the best aided condition to compare.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 4
Percentage of participants | 75 [19 to 99]

ADVERSE EVENTS:
Description: Death, serious adverse events and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Nucleus CI532 Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will be able to publish and/or present their own data. The publishing investigator will provide the sponsor with a manuscript copy of the abstract and paper at least 30 days in advance of publication or presentation. If the publication contains information that the sponsor at his discretion finds worth protecting in the form of a patent or trademark etc., the sponsor has the right to delay the publication or presentation for 90 days.

DOCUMENTS (2):
  • Study Protocol (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03039283/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03039283/SAP_001.pdf